CLINICAL TRIAL: NCT05734885
Title: The Effect of Partner Massage in Labor on Pain, Anxiety and Birth Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ayse Nur Atas, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0000-0003-3096-3599
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Midwifery; Labor Delivery; Massage
Keywords: Labor; massage; partner massage; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The sample size of the study was calculated based on the results of a study aiming to determine the effect of birth dance applied with the support of a spouse and midwife during labor on birth pain and satisfaction [19]. It was found as 116 participants, including 39 in each group, on the G*power 3.1.9.2 (Ver. 3.1.9.2) [20] software, based on an effect size of 0.71, a power of 0.95, and an alpha level of 0.05. Considering some attrition, an additional 15% was added to the sample size, and the study was planned to be conducted with 141 women (47 in the partner massage group, 47 in the midwife massage group, and 47 in the control group). During monitoring, two participants were lost from each group. Eventually, the study was completed with a total of 135 women, 45 in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midwife Massage Experimental Group (1) (Experimental): Back and sacral massage will be applied to pregnant women in labor in the application group. Massage will be applied by the research midwife. Midwife massage will be performed when cervical dilation is 5-6 cm and 8-9 cm.
  Massage application time will last 20 minutes.
  Interventions: Other: Back and Sacral massage massage application
- Spouse Massage Experimental Group (2) (Experimental): Back and sacral massage will be applied to pregnant women in labor in the application group. Massage will be applied by the spouse of the pregnant woman. Massage will be performed when cervical dilation is 5-6 cm and 8-9 cm.
  Massage application time will last 20 minutes.
  Interventions: Other: Back and Sacral massage massage application
- Control Group (No Intervention): It will be perform routine practice who the women in the control group.

INTERVENTIONS:
Other: Back and Sacral massage massage application — Massage will be applied to the pregnant woman in the position preferred by the pregnant woman. Circular movements are applied to the sacrum with the thumb. Pressure is applied to both sides of the spinal cord with the thumb. The thumb is moved towards the hip of the pregnant woman at 1.5 cm intervals, starting from the lower part of the pelvis and the sacrum. The palm is placed in direct contact with the mother's sacrum and pressure is applıed. The massage is completed by making a bunch of flowers from the sacrum upwards, towards the shoulder and around it.
  Arms: Midwife Massage Experimental Group (1); Spouse Massage Experimental Group (2)

SUMMARY:
H1-1 = There will be a difference between the pain levels of the partner massage group, midwife massage group, and control group following the massage application.

H1-2 = There will be a difference between the state anxiety levels of the partner massage group, midwife massage group, and control group following the massage application.

H1-3 = There will be a difference between the active phase durations of the partner massage group, midwife massage group, and control group following the massage application.

DETAILED DESCRIPTION:
Supporting the woman with massage during the labor process reduces the severity of pain, provides general relaxation and reduces anxiety. The application of spousal massage for supportive care to the woman during the labor process can provide important positive results in terms of providing both physical and emotional support. A positive perception of birth can be strengthened by meeting women's needs at a higher level. This may contribute to effective pain management, reduction of anxiety in women, improvement of birth outcomes and positive neonatal health outcomes. When the literature is examined, it has been determined that the scope and number of studies examining the effect of partner massage in labor on pain, anxiety and birth process is very limited, and there is no study on the subject in the national literature.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 20-35
* Term pregnancies (those at 37-41 weeks of gestation)
* Those with a single fetus
* Primiparous
* Those who do not have any risk factors during pregnancy (Preeclampsia, premature rupture of membranes, placental anomalies, macrosomic baby, etc.)
* Those who do not have any chronic disease
* Pregnant women who do not have skin disease, infection or varicose affecting the massage application.
* Pregnant women with no deterioration in skin integrity
* Those with cervical dilatation less than 4 cm
* Those who are open to communication, mentally and mentally healthy
* Those who agreed to participate in the study
* Pregnant women with a spouse who agree to apply and apply massage for the spouse/partner massage group.

Exclusion Criteria:

* Those who are in the active and transitional phase of labor
* Abnormal changes in fetal heartbeats
* Unexpected complication in pregnancy and fetus
* Pregnant women who use pharmacological methods to reduce pain during labor
* Pregnant women with contraindications for massage application (deterioration of skin integrity, varicose veins, skin disease and infection)
* Pregnant women who are reluctant to continue participating in the research

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 135 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Pregnant Introduction Form | in active phase on labor (4 cm and less vaginal dilatation)
  The pregnancy information form, which was prepared by the researcher following a literature review, consisted of 18 questions about some socio-demographic characteristics of pregnant women (age, education level, social security status, etc.) and their obstetric characteristics (gestational week, problems during pregnancy, etc.),
Labor Monitoring Form | in labor and in the first 24 hours postpartum
  This form was developed by the researcher following a literature review. It consisted of five items about the practices applied to pregnant women during labor (interventions applied during labor (forceps, vacuum, etc.)) and the characteristics of the newborn in the postpartum period (Apgar score, newborn weight, etc.),
Partograph | in active phase on labor (4, 5-6, 8-9 cm vaginal dilatation)
  This is a tool used to assess the progress of labor and the health status of the fetus. It is used from the active phase of labor. It visualizes the progress of labor; cervical dilatation, the level of the fetal head, the frequency and duration of uterine contractions, fetal heart rate, the presence of amniotic membrane, and the color of amniotic fluid are evaluated and recorded on a graph paper Its central feature is a graph used to record the progress of cervical dilation, as determined by vaginal examination.
  Indicators are plotted on the graph each time they are checked:
  * Maternal indicators:
    * Time of spontaneous or artificial rupture of the membranes
    * Uterine contractions (number per 10 minutes and duration)
    * Drugs administered (oxytocin, antibiotics, etc.)
  * Foetal indicators:
    * Foetal heart rate
    * Amniotic fluid (colour, odour and quantity)
    * Descent of the foetal head and head moulding
Visual Analog Skala-VAS | in active phase on labor (4, 5-6, 8-9 cm vaginal dilatation)
  The VAS was first developed by Price et al. (1983). The VAS is used to measure perceived pain. 10 cm, which says painlessness at one end and the most severe pain at the other end. On a (100 mm.) ruler, the patient describes his or her pain by drawing a line, pointing, or pointing. The length of the distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found shows the severity of the patient's pain.
Spielberger State Anxiety Scale | in active phase on labor (4, 5-6, 8-9 cm vaginal dilatation)
  It was developed by Spielberg et al in 1970. It was adapted into Turkish by Öner and Le Compte in 1983 (Öner & Le Compte, 1983; Özusta, 1995). The state anxiety scale is a scale that determines how an individual feels at a particular moment and situation. It requires the individual to answer the feelings or behaviors he/she experiences in his/her situation by marking one of the options such as (1) Not at all, (2) A little, (3) A lot and (4) Completely. The state anxiety scale consists of 20 statements. The score obtained from the scale can vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety. In the scoring made in accordance with the criteria directive, 0-19 points are evaluated as "absent", 20-39 points as "mild", 40-59 points as "moderate", 60-79 points as "severe" and 80 points as severe anxiety (Dönmez, Yeniel, & Kavlak, 2014).
Assessment of Satisfaction Scale | in the first 24 hours postpartum
  This scale was adopted by the researcher from the "Visual Analog Scale (VAS)", which individuals can easily understand [35]. The VAS helps measure some variables numerically, which is not possible otherwise. This scale was used to evaluate the satisfaction of the women in the study group with the massage application and the labor process. The numbers between 0 and 10, which were intended to indicate the point corresponding to the satisfaction status, were placed on a vertical line. A score of 0 on the scale indicated "not satisfied at all", while a score of 10 indicated "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Nur Ataş, Principal Investigator — Necmettin Erbakan University, Faculty of Medicine
Locations (1):
- Ayşe Nur Ataş, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No